CLINICAL TRIAL: NCT00628316
Title: Effects of Caffeine Consumption on Tinnitus Perception
Brief Title: Effects of Caffeine in Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Medicina de Valenca (Other)
Responsible Party: Ricardo Rodrigues Figueiredo, MD, MSc, University of Valencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMV 001 2008
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2008-02

CONDITIONS: Tinnitus
Keywords: tinnitus; caffeine
MeSH Terms: conditions — Tinnitus | interventions — Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: caffeine — caffeine daily intake will be reduced form 150 ml per day

SUMMARY:
Caffeine intake is reported by many authors to enhance the perception of tinnitus. The aim of this study is to determine the effects of 1 month caffeine intake reduction in the scores of validated questionnaire Tinnitus Handicap Inventory (THI) and in a visual-analog scale (VAS).

DETAILED DESCRIPTION:
A group of 50 patients who takes more than 3 small cups (50 ml) of caffeine daily and have tinnitus will be asked to reduce caffeine intake for 1 month. Scores of THI and VAS will be taken before and after this period.

ELIGIBILITY:
Inclusion Criteria:

* tinnitus for more than 6 months
* THI > 38
* no central acting drugs in the last 6 months
* tympanogram type A-n
* daily intake of caffeine greater than 150 ml

Exclusion Criteria:

* vascular and muscular tinnitus
* concomitant TMJ disorders
* abnormal otoscopy
* mixed and conductive hearing losses
* Ménière disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory | 30 days

SECONDARY OUTCOMES:
Visual Analog Scale | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo R Figueiredo, MD,MSc, Study Chair — Faculdade de Medicina de Valença
Locations (2):
- Brazil (2):
  - Faculdade de Medicina de Valença, Valença, Rio de Janeiro
  - OTOSUL Otorrinolaringologia Sul-Fluminense, Volta Redonda, Rio de Janeiro